CLINICAL TRIAL: NCT02155673
Title: A Phase 2 Extension Study of Study GCS-100-CS-4002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCS-100-CS-4003
Record Dates: First submitted 2014-04-09; First posted 2014-06-04 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — GCS-100

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dose GCS-100 (Experimental): Low dose of GCS-100
  Interventions: Drug: GCS-100
- High Dose GCS-100 (Experimental): GCS-100 High dose
  Interventions: Drug: GCS-100

INTERVENTIONS:
Drug: GCS-100 — 1.5 mg/m2 or 30 mg/m2 GCS-100. GCS-100 will be administered as IV infusions once weekly for 8 weeks with a 1 week and 4 week follow-up period and then at least every 30 days for up to a total of 1 year.

SUMMARY:
The primary objective of this study is to determine the safety and tolerability of extended dosing of GCS-100 in patients with CKD.

DETAILED DESCRIPTION:
Galectin-3 contributes to fibrosis, is elevated in patients with ESRD, and correlates with adverse outcomes. Animal models with genetic knockout of galectin-3 demonstrate a reduction in structural and functional deficits in the kidney. GCS-100 is a galectin-3 antagonist that has been shown to reduce fibrosis pre-clinically. Based on the role of galectin-3 and fibrosis in kidney disease, the Sponsor believes GCS-100 may be effective at treating patients with CKD.

Study GCS-100-CS-4002 is an ongoing randomized, placebo controlled study of GCS-100 in Stage 3b and 4 CKD. The objective of the study is to determine the safety and efficacy of 8 weekly injections of GCS-100 on eGFR. Patients who have completed that study without adverse safety events, may be asked to participate in this study to test the safety of prolonged administration of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is capable of understanding the purpose and risks of the study and is able to provide written informed consent
2. Subject was enrolled in and completed the End of Study (Day 85) of GCS-100-CS-4002

Exclusion Criteria:

1. Subject experienced a Grade 3 or worse adverse event related to GCS-100 in clinical study GCS-100-CS-4002
2. Systolic blood pressure ≤90 mmHg and ≥160 mmHg and diastolic blood pressure ≤40 mmHg and ≤100 mmHg at screening
3. Subject has clinical laboratory results of:

   1. Hemoglobin: ≤9g/dL
   2. Total bilirubin: >1.5X the upper limit of normal (ULN)
   3. ALT and/or AST: >2.5X ULN
4. Subject has a concomitant disease or condition, including laboratory abnormalities, which, in the opinion of the investigator, could interfere with the conduct of the study or put the subject at unacceptable risk
5. Subject who may require renal replacement therapy within the next 2 months, at the discretion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of Safety | Participants will be followed for the duration of the study, up to 1 year with a four week additional follow-up period.
  Evaluation of safety measures for long-term dosing including collection of adverse events in clinically significant changes in lab values

CONTACTS AND LOCATIONS:
Overall Officials: George Tidmarsh, MD, PhD, Study Director
Locations (5):
- United States (5):
  - Southwest Clinical Research Institute, LLC, Tempe, Arizona
  - California Institute of Renal Research, La Mesa, California
  - Denver Nephrology, Denver, Colorado
  - Mountain Kidney and Hypertension Associates, PA, Asheville, North Carolina
  - Clinical Advancement Center, PLLC, San Antonio, Texas